CLINICAL TRIAL: NCT03158987
Title: Regional Differences in Human Immunodeficiency Virus (HIV) Testing Procedures in Eastern German Federal States
Brief Title: Regional Differences in Human Immunodeficiency Virus (HIV) Testing
Acronym: HIVRegional
Status: Completed | Type: Observational
Sponsor: Jena University Hospital (Other)
Collaborators: University of Magdeburg (Other); University of Leipzig (Other); University of Rostock (Other); Technische Universität Dresden (Other); MUC Research GmbH (Other)
Responsible Party: Sponsor
Other Study IDs: ZKS00
Record Dates: First submitted 2017-05-17; First posted 2017-05-18 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2017-05

CONDITIONS: HIV Seropositivity; CD4+ T Lymphocytopenia
MeSH Terms: conditions — HIV Seropositivity; T-Lymphocytopenia, Idiopathic CD4-Positive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical record review — Review of medical records of patients diagnosed for the first time as HIV seropositivity

SUMMARY:
This retrospective observational study aims at the examination of regional differences in the procedure of referral for serological HIV testing between eastern (new) and western (old) German federal states.

DETAILED DESCRIPTION:
Increasing incidence of HIV infections urges early recognition and timely introduction of therapy. Regional differences in referral approach and patient behavior are presumably associated with considerable delays in infection recognition and therapy onset. Comparison of records of new cases which were diagnosed in 2014 in several eastern federal states and a major western German city is expected to disclose whether the regionally preferred type of the primary care institution affects the time point of first diagnosis and the elapsed time since the emergence of the infection, as assessed by Cluster of Differentiation 4 positive (CD4+) lymphocyte counts and manifestation of clinical symptoms of immune deficiency.

ELIGIBILITY:
Inclusion Criteria:

* first-time HIV seropositivity

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have displayed for the first time a serological proof of HIV infection
Sampling Method: Probability Sample
Enrollment: 999 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Type of HIV-verifying medical institution | 1 day
  Medical Institution (university hospital, general practitioner, specialized medical office) which has diagnosed HIV seropositivity for the first time

SECONDARY OUTCOMES:
CD4+ lymphocyte counts | 1 day
  Number of CD4+ lymphocytes at the time of HIV diagnosis
Symptoms of AIDS-related diseases | 1 day
  Presence of AIDS-related disease symptoms at the time of first HIV seropositivity diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Schleenvoigt, M.D., Study Director — University Hospital Jena
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No